CLINICAL TRIAL: NCT06537622
Title: Implementation of Best Practices for Early Diagnosis of Cerebral Palsy (CP) in Very Preterm Infants: a Stepped-wedge Cluster Randomized Controlled Trial (RCT)
Brief Title: Best Practices Fo Early Diagnosis of Cerebral Palsy
Acronym: CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: IWK Health Centre (Other); St. Boniface Hospital (Other); Sunnybrook Health Sciences Centre (Other); Montreal Children's Hospital of the MUHC (Other); Harvard University (Other); University of British Columbia (Other); Queen Alexandra Centre for Children's Health, Victoria (Unknown); Jewish General Hospital (Other); CHU de Quebec-Universite Laval (Other); BC Women's Hospital & Health Centre (Other); Dr. Everett Chalmers Hospital (Unknown); Janeway Children's Health and Rehabilitation Centre (Unknown); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Horizon Health Network (Other); Moncton hospital (Unknown); Windsor Regional Hospital (Other); Maisonneuve-Rosemont Hospital (Other); The Hospital for Sick Children (Other); MOUNT SINAI HOSPITAL (Other); Health Sciences Centre, Winnipeg, Manitoba (Other); Glenrose Foundation (Other); Hamilton Health Sciences Centre (Unknown); London Health Sciences Centre (Other); Children's Hospital of Eastern Ontario (Other); Kingston Health Sciences Centre (Other); Foothills Medical Centre (Other); Island Health, Victoria, BC (Other); Canadian Premature babies Foundation (Unknown)
Responsible Party: Principal Investigator, Thuy Mai Luu, Pediatrician, researcher and Medical director of the Canadian Neonatal Follow-up Network (CNFUN), St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MP-21-2024-7044
Record Dates: First submitted 2024-07-10; First posted 2024-08-05 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy; Prematurity
Keywords: Corrected age; very preterm infants; Developmental functioning; Guideline; Diagnosis; Randomized controlled trial
MeSH Terms: conditions — Cerebral Palsy; Premature Birth; Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: CNFUN sites are the unit of randomization to the order in which they receive the implementation strategy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention aim (Other): To assess the effectiveness of the clinical practice guideline - cerebral palsy detecting early signs of CP at a younger age. More specifically, to reduce the age at detecting early signs of CP from an estimated CA of 11 months (prior to CPG-CP implementation) to 8 months. To determine whether using both the general movement assessment and Hammersmith infant neurological examination is more performant than the HINE alone in identifying early signs of CP. To examine if CPG-CP implementation is associated with better developmental functioning at 18-24 months CA.
  Interventions: Other: Implementation group
- Implementation aim (Other): Using the RE-AIM framework : To assess REAch of the intervention strategies to the target audience of clinicians in CNFUN programs.To assess Implementation fidelity to the CPG-CP and the implementation strategies. To assess Maintenance of the CPG-CP over time.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Implementation group — Implementation strategies to increase uptake of the clinical practice guidelines for earlier diagnosis of cerebral palsy
  Arms: Intervention aim
Other: Standard of care — No active implementation strategies
  Arms: Implementation aim

SUMMARY:
In this research, the investigators are using an implementation science approach to enhance the uptake of a clinical practice guideline for earlier diagnosis of cerebral palsy (i.e. what is being implemented) in neonatal follow-up clinics across Canada. This clinical practice guideline should be part of what neonatal follow-up specialists do in their routine clinical work with children born preterm. However, there is a wide variability in practice. The goal of this project is to harmonize practices in the neonatal follow-up community in agreement with international recommendations for earlier diagnosis of cerebral palsy. This research will measure if clinicians are truly following the clinical practice guideline. If not, implementation strategies that address barriers and leverage on facilitators will be deployed for successful uptake of the clinical practice guideline. This research will also assess whether implementation of the clinical practice guideline is associated with better patient outcomes.

DETAILED DESCRIPTION:
Children born preterm have an increased risk for brain-based disabilities, including cerebral palsy (CP), with lower gestational age (GA) incurring higher vulnerability. The rate of CP in very preterm children born before 29 weeks' GA is 6.1%.The 2017 international recommendations for Early, accurate diagnosis and early intervention in CP provides an evidence-based approach for prompt referral to targeted services to optimize child outcomes. Early diagnosis and intervention during the optimal window of brain plasticity has the potential to improve developmental functioning. Best practice guidelines also exist on how to convey an early diagnosis of CP in a compassionate way, as poor communication can affect parental mental health. The Canadian Neonatal Follow-Up Network (CNFUN) has partnered with the parent-led Canadian Premature Babies Foundation (CPBF) and key stakeholders to adapt these clinical practice guidelines to the Canadian context (CPG-CP). These CPG-CP promote the use of the General Movement Assessment (GMA) and the Hammersmith Infant Neurological Examination (HINE) for identification of early signs of CP. The CPG-CP also propose clinical care pathways and an approach for communicating findings. The overall goal of the CPG-CP is to improve clinicians' ability to accurately recognize the earliest signs of CP that warrant immediate actions (as opposed to a wait-and-see approach). Using a hybrid effectiveness-implementation trial design, the investigators will assess whether the implementation strategy is successful in increasing the uptake of the CPG-CP by CNFUN programs. Concurrently, the investigators will test the effectiveness of implementing the CPG-CP in detecting early signs of CP at a younger age in preterm infants born <29 weeks' GA. The investigators will secondarily compare whether using both the GMA and HINE is more performant than the HINE alone in identifying early signs of CP. Finally, the investigators will examine whether developmental functioning at 18-24 months corrected age (CA) improves after CPG-CP implementation.

This proposal aims to reduce the gap in care related to the early identification of CP in children born very preterm across Canada. Using a hybrid effectiveness-implementation study design, the investigators will implement the CPG-CP in the real-world setting of CNFUN sites, to improve clinicians' ability to detect the early signs of CP in very preterm infants. Early diagnosis enables the initiation of targeted interventions and engagement of support services. Harnessing neuroplasticity through early and specific therapy can improve children's overall development and functioning. The effectiveness of the CPG-CP on improving clinical outcomes relies on a successful implementation process that considers the interplay between inner (i.e., within neonatal follow-up programs), outer (e.g., local health care system), and individual patient and clinician characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Infants born preterm at less than 29 weeks' GA and their parents
* Admission to a Neonatal Intensive Care Unit (NICU) participating in the Canadian Neonatal Network (CNN).

Exclusion Criteria:

* Death prior to first visit in clinic
* Major congenital malformation and/or significant chromosomal defects affecting development beyond preterm birth
* Child moved outside Canada prior to first visit in clinic.

Ages: 2 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Intervention : corrected age at detection of early signs of CP. | Birth to 18-24 months CA
  This is calculated from the date at which the clinician identifies early signs of CP and shares this diagnosis with family. This diagnosis must be followed by an immediate action i.e., referral for CP-targeted intervention and/or evaluation. Outcome data will be collected through retrospective chart review.
Intervention : Developmental functioning at 18-24 month CA | Birth to 18-24 months CA
  Evaluation of the developmental functioning using the Bayley Scales of Infant and Toddler Development, 4th edition (Bayley-4), a widely used, standardized, norm-referenced instrument for direct assessment of children aged 1-42 mo. Cognition, language, and motor composite scores are obtained (mean 100±15).

SECONDARY OUTCOMES:
Implementation : RE-AIM framework - Reach, Effectiveness, Adoption | Up to 48 months
  Reach of the intervention strategies to the target audience of clinicians participating in the CNFUN.
Implementation : RE-AIM framework - Implementation | Up to 48 months
  Implementation fidelity to the CPG-CP and the implementation strategies.
Implementation : RE-AIM framework - Maintenance | Up to 48 months
  Maintenance of the practice of CPG-CP over time.

CONTACTS AND LOCATIONS:
Overall Officials: Luu Thuy Mai, MD, M.Sc., Principal Investigator — CHU Sainte-Justine hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will not be available for sharing. Only aggregated data can be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will be sharing this material starting in January 2025 as soon as ethics approval has been obtained from all sites until the end of the study.
Access Criteria: The individual is affiliated with a non-profit organization or a university-based research institution.
URL: https://canadianneonatalfollowup.ca/data-request/